CLINICAL TRIAL: NCT05093335
Title: In-human CXCR4 Imaging of Hematologic and Solid Tumors Using [68Ga]-Pentixafor-PET
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-356
Record Dates: First submitted 2021-10-01; First posted 2021-10-26 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Non-Hodgkin Lymphoma; Multiple Myeloma; Histiocytic Neoplasms; Erdheim-Chester Disease; Rosai-Dorfman Disease
Keywords: [68Ga]-Pentixafor; PET/CT scan; In-human CXCR4 Imaging; 21-356; Symptomatic multiple myeloma; pre-cursor myeloma; MGUS; SMM; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Multiple Myeloma; Erdheim-Chester Disease; Histiocytosis, Sinus | interventions — 68Ga-pentixafor

STUDY DESIGN:
Intervention Model Description: This protocol is a pilot protocol.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- [68Ga]-Pentixafor (Experimental): An intravenous bolus of 3 -5 mCi [68Ga]-Pentixafor will be injected in all participants that will be imaged on a hybrid PET/CT device. Any of the following factors may determine if imaging cannot be performed: tolerance/compliance in the PET/CT scanner; dose availability; dose quality control; availability of the PET/CT scanner or availability of study personnel. [68Ga]-Pentixafor uptake dynamics / pharmacokinetics will be evaluated by PET/CT performed with a low-dose CT component used for PET attenuation correction (1-2 mSv). [68Ga]-Pentixafor-PET/CT scan duration will be approximately 1.5 hours. Some patients will have two scans.
  Interventions: Drug: [68Ga]-Pentixafor

INTERVENTIONS:
Drug: [68Ga]-Pentixafor — An intravenous bolus of 3 -5 mCi of [68Ga]-Pentixafor will be injected in all participants.

SUMMARY:
The purpose of this study is to determine the uptake of the imaging agent [68Ga]-pentixafor with PET/CT scans in people with monoclonal gammopathy of undetermined significance (MGUS), smoldering multiple myeloma (SMM), and non-Hodgkin lymphoma (NHL), or you have histiocytic neoplasms (Langerhans cell histiocytosis (LCH), Erdheim-Chester disease (ECD) and/or Rosai-Dorfman disease (RDD).

ELIGIBILITY:
Inclusion Criteria:

Twenty patients with histologically proven treatment-naïve, therapy-refractory or relapsed blood cancers meeting the below criteria will be included:

* Indolent B- or T-cell Non-Hodgkin lymphoma (including cutaneous lymphomas) or Non-Hodgkin lymphoma with variable FDG uptake and clinical course, such as mantle cell lymphoma; and measurable disease according to Lugano criteria

or

* Histiocytic neoplasms (Langerhans cell histiocytosis (LCH), Erdheim-Chester disease (ECD) and/or Rosai-Dorfman disease (RDD)
* MGUS/SMM or MM according to IMWG definitions
* Solid tumors, such as lung cancers, meningioma, adrenocortical neoplasms including cortisol-producing adenomas or high suspicion for tumor, such as in patients with Cushing's disease.
* Age ≥18
* Negative serum pregnancy test for female volunteers of childbearing age and potential (as defined by MSKCC Standards & Guidelines) from assays obtained <2 weeks prior to study enrollment/intervention; or negative urine pregnancy test performed on the day of intervention
* MSKCC patients

Exclusion Criteria:

* Breast-feeding
* History of renal functional disorders (chronic kidney disease with eGFR<30)
* Refusal or inability to tolerate the scanning procedure (e.g., due to claustrophobia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Tumor standard uptake value (SUV) | 1 year
  Means and 95% confidence intervals for [68Ga]-Pentixafor standardized uptake values (SUV) and tumor-to-background ratios (TBR) of tumors will be recorded. Uptake will be measured in tumors.

CONTACTS AND LOCATIONS:
Overall Officials: Anton Nosov, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm